CLINICAL TRIAL: NCT03935321
Title: Antibodies Against Nogo-A to Enhance Plasticity, Regeneration and Functional Recovery After Spinal Cord Injury - A Multicenter International Randomized Double Blind Placebo Controlled Phase II Clinical Proof of Concept Trial
Brief Title: NISCI - Nogo Inhibition in Spinal Cord Injury
Acronym: NISCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: EMSCI.org (Unknown); State Secretariat for Education Research and Innovation, Switzerland (Other); Horizon 2020 - European Commission (Other); Foundation Wings For Life (Other); Swiss Paraplegic Research, Nottwil (Network); Heidelberg University Hospital Spinal Cord Injury Center (Unknown); KKS Netzwerk (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT No. 2016-001227-31
Record Dates: First submitted 2019-03-25; First posted 2019-05-02 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injury, Acute
Keywords: Tetraplegia; Trauma; Upper limbs function
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with acute cervical spinal cord injury: NG-101 (Active Comparator)
  Interventions: Drug: NG-101
- Patients with acute cervical spinal cord injury: Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: NG-101 — 6 intrathecal bolus injections, each of 45mg
  Arms: Patients with acute cervical spinal cord injury: NG-101
Drug: Placebos — 6 intrathecal bolus injections, each of 45mg
  Arms: Patients with acute cervical spinal cord injury: Placebo

SUMMARY:
The purpose of the NISCI trial is to test if an antibody therapy can improve movement and quality of life of tetraplegic patients. A previous trial showed this treatment is safe and well accepted. This is a placebo controlled, randomized, double blind, multicenter, multinational study to assess the safety, tolerability, feasibility and preliminary efficacy of early (within 4-28 days post injury) initiation of treatment with repeated bolus injections of NG-101 in cervical acute SCI patients. The study has 3 phases: screening/baseline Phase, treatment phase, and a follow-up phase.

The study design will allow simultaneous enrolment of patients with complete or incomplete SCI. Enrolment and stratification of the patients is based and individualized prediction of upper limb outcomes.

For further information please visit NISCI website: https://nisci-2020.eu

ELIGIBILITY:
Inclusion Criteria:

* Acute cervical spinal cord injury (SCI) (Neurological level of injury C1-C8 with confirmed classification of ASIA impairment scale (AIS) A-D at screening and predicted upper extremities motor score (UEMS) recovery of less than 41/50 (according to the URP prediction model)
* 4-28 days post-injury
* No required mechanical ventilation or patients that not completely depend on mechanical ventilation
* Hemodynamically and clinical stable patient according to the acute SCI condition at baseline
* Written informed consent
* Cooperation and willingness to complete all aspects of the study
* Ability of subject to understand character and individual consequences of the study

Exclusion Criteria:

* Complete anatomical transection confirmed by magnetic resonance imaging (MRI)
* Trauma caused by ballistic or other injury that directly penetrates the spinal cord including gunshot and knife wounds
* Major brachial or lumbar plexus damage/trauma
* Significant head trauma or other injury that was, in the opinion of the investigator, sufficient to interfere with the assessment of the spinal cord function
* Other significant pre-existing or current severe systemic disease such as lung, liver (exception: history of uncomplicated Hepatitis A), gastorintestinal, cardiac, immunodeficiency (including anamnestic known HIV) or kidney disease; or active malignancy
* History of or an acute episode of Guillain-Barre syndrome
* History of recent (6 months) meningitis or meningoencephalitis
* History of refractory epilepsy
* History of or current autoimmune disease
* Patients with uncontrolled bleeding diathesis and/or who require concomitant treatment with coumarin anticoagulant
* Presence of any unstable medical or psychiatric condition
* Drug dependence any time during the 6 month's preceding study entry
* Pregnant or nursing women
* History of a life-threatening allergic or immune mediated reaction
* Patients with the presence of infection around the location where the spinal needle insertions are planned for applying the intrathecal injections
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulations
* Patients who are unconscious
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Change of upper extremity motor scores (UEMS) according to the International Standards for the Neurological Classification of Spinal Cord Injury | Change from screening at day 168

SECONDARY OUTCOMES:
Change of effect on motor and sensory function according to the ISNCSCI protocol | Change from screening at day 168
Change of effect on autonomic dysfunction measured by bladder diary | Change from screening at day 168
Change of effect on quality life of patients with neuro-urological disorders as measured by Qualiveen questionnaire | Change from screening at day 168
Change of effect on autonomic dysfunction as measured by bladder function assessment | Change from screening at day 168
Change of effect on functioning, evaluated by the Spinal Cord Independence Measure (SCIM-III) | Change from baseline at day 168
Change of effect on hand/upper limb function as assessed by the Graded and Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) | Change from baseline at day 168
Change of effect on the Walking Index for Spinal Cord Injury (WISCI | Change from baseline at day 168
Change of effect on 10 meter walk test (10mWT) | Change from baseline at day 168
Change of effect on 6-minute walking test (6MWT) | Change from baseline at day 168
Change of effects on nerve conducting velocity | Change from screening at day 168
Change of effects on somatosensory evoked potentials | Change from screening at day 168
Evaluation of concentration NG-101 in serum (pharmacokinetics) | Change from day 0 at day 84
Evaluation of concentration NG-101 in CSF (pharmacokinetics) | Change from day 0 at day 84

CONTACTS AND LOCATIONS:
Overall Officials: Armin Curt, Prof., Principal Investigator — Universität Zürich / University Hospital Balgrist; Norbert Weidner, Prof., Principal Investigator — University Hospital Heidelberg
Locations (13):
- Spinal Cord Unit, University Hospital Motol, Prague, Czechia
- Germany (8):
  - Klinik für Querschnittgelähmte, Klinikum Bayreuth, Bayreuth
  - Behandlungszentrum für Rückenmarkverletzte, Unfallkrankenhaus Berlin, Berlin
  - Abteilung für Rückenmarkverletzte, BG Universitätsklinikum Bergmannsheil gGmbH, Bochum
  - Zentrum für Rückenmarkverletzte und Klinik für Orthopädie, BG Klinikum Bergmannstrost, Halle
  - Klinik für Paraplegiologie, Universitätsklinikum Heidelberg, Heidelberg
  - Zentrum für Tetra- und Paraplegie, Orthopädische Klinik Hessisch Lichtenau gGmbH, Hessisch Lichtenau
  - Zentrum für Rückenmarksverletzte, Unfallklinik Murnau, Murnau am Staffelsee
  - BG Klinik Tübingen, Tübingen
- Center for Neurorehabilitation, Fundacio Institut Guttmann, Barcelona, Spain
- Switzerland (3):
  - Rehab Basel, Basel
  - Schweizer Paraplegikerzentrum, Nottwil
  - Universitätsklinik Balgrist, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kucher K, Johns D, Maier D, Abel R, Badke A, Baron H, Thietje R, Casha S, Meindl R, Gomez-Mancilla B, Pfister C, Rupp R, Weidner N, Mir A, Schwab ME, Curt A. First-in-Man Intrathecal Application of Neurite Growth-Promoting Anti-Nogo-A Antibodies in Acute Spinal Cord Injury. Neurorehabil Neural Repair. 2018 Jun;32(6-7):578-589. doi: 10.1177/1545968318776371. Epub 2018 Jun 5. PMID 29869587
- [Derived] Giagiozis M, Lerch I, Linke AD, Jutzeler CR, Rupp R, Abel R, Benito-Penalva J, Waldmann J, Maier D, Baumberger M, Kriz J, Badke A, Hund-Georgiadis M, Weidner N, Demko L, Curt A. Feasibility and Sensitivity of Wearable Sensors for Daily Activity Monitoring in Spinal Cord Injury Trials. Neurorehabil Neural Repair. 2025 Oct;39(10):814-825. doi: 10.1177/15459683251352556. Epub 2025 Jul 10. PMID 40637209
- [Derived] Weidner N, Abel R, Maier D, Rohl K, Rohrich F, Baumberger M, Hund-Georgiadis M, Saur M, Benito J, Rehahn K, Aach M, Badke A, Kriz J, Barkovits K, Killeen T, Farner L, Seif M, Hubli M, Marcus K, Maurer MA, Robert B, Rupp R, Scheuren PS, Schubert M, Schuld C, Sina C, Steiner B, Weis T, Hug A, Bolliger M, Weiskopf N, Freund P, Hothorn T, Schwab ME, Curt A; Nogo Inhibition in Spinal Cord Injury Study Group. Safety and efficacy of intrathecal antibodies to Nogo-A in patients with acute cervical spinal cord injury: a randomised, double-blind, multicentre, placebo-controlled, phase 2b trial. Lancet Neurol. 2025 Jan;24(1):42-53. doi: 10.1016/S1474-4422(24)00447-2. PMID 39706632